CLINICAL TRIAL: NCT06843785
Title: Effects of Two Different Squat Exercise Patterns on Muscle Strength, Performance, Low Back Pain and Balance in Young Adult Healthy Individuals
Brief Title: Comparison of the Effectiveness of Two Different Squat Exercises in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Uskudar23
Record Dates: First submitted 2025-02-19; First posted 2025-02-25 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Balance; Distorted; Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- knee past toes squat (Experimental): A squatting program with the desired characteristics will be applied
  Interventions: Other: Squat with knees over toes
- control (Active Comparator): no intervention will be applied
  Interventions: Other: control
- knee not past toes squat (Experimental): A squatting program with the desired characteristics will be applied
  Interventions: Other: Squat where the knee does not pass the toes

INTERVENTIONS:
Other: Squat with knees over toes — Participants are instructed to stand comfortably with feet pelvis-width apart and approximately 15-30° to the side with arms extended in front of them. Participants are asked to squat to their most comfortable point, looking straight ahead, without heels leaving the floor, and to hold the position for 2 seconds before returning to the original standing position. The distance between the hips and the floor is measured vertically using a ruler for squat depth. Three trials are performed and the average of the three trials is used for further analysis.
  Arms: knee past toes squat
Other: Squat where the knee does not pass the toes — In the limited squat exercise, the position of the most anterior part of the knee is not allowed to extend beyond the toes. In the limited squat exercise, a wooden board is placed just distal to the first toe of each foot, and the 60 cm wide wooden board restricts knee movement. Participants are instructed to stand comfortably with their feet pelvis-width apart and approximately 15-30° to the side, and their arms extended in front of them. Participants are asked to squat to 90° of knee flexion, looking straight ahead, without the heels leaving the floor, and to hold the position for 2 seconds, then return to the original standing position. Squat depth is determined by measuring 90° of knee flexion using a goniometer placed on the knee and measured vertically between the hip and the floor using a ruler. Three trials are performed, and the average of the three trials is used for further analysis.
  Arms: knee not past toes squat
Other: control — Participants will not be subjected to any intervention and will not be asked to perform any action.
  Arms: control

SUMMARY:
The aim of our study is to compare the effects of two different squatting patterns, with and without the knees passing the toes, on low back pain, muscle strength and balance.

DETAILED DESCRIPTION:
A total of 60 volunteer participants between the ages of 18-30, who are in the active category of the International Physical Activity Assessment Questionnaire Short Form, are planned to be included in the study. Individuals participating in the study will be divided into 3 groups using a computer randomization system and a closed envelope method. Group I (n=20); squatting with the knees passing the toes (PI), Group II (n=20); squatting with the knees not passing the toes (PG) and Group III (n=20); control group (CG). Squatting with the knees passing the toes (PI); squatting with the knees not passing the toes (PG) will be applied to the study groups as a home program for 4 weeks and will be checked with an exercise diary. Participants will be re-evaluated at the end of the exercise program. No training program will be applied to the control group and they will be asked to continue their daily lives and participants will be evaluated at 4-week intervals. The training program of 1 set; 20 repetitions; 30 seconds active contraction/30 seconds rest is applied to the PI and PG groups 3 days a week, every other day for 6 weeks. The training program of the groups is monitored by a physiotherapist for 6 weeks via telerehabilitation technologies. All participants will be evaluated for back pain, knee pain, muscle thickness, muscle strength, function and balance before and at the end of the program and the data obtained will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-30,
* According to International Physical Activity Questionnaire - Short Form Being physically active
* Not having any psychological, neurological, orthopedic and rheumatic disorders,
* Not having a history of fractures or surgeries affecting the lower extremities in the last year,
* Being able to do at least one traditional squat exercise
* Being able to communicate in Turkish (written and verbal) Exclusion criteria
* Being pregnant or suspected of being pregnant
* Knee valgus diagnosis
* Pes planus or pes cavus diagnosis in the foot
* Hip rotation diagnosis
* Strength deficit between two extremities
* A history of acute osteoarthritis in the knee
* Regular medication use or use of NSAIDs and similar disease-modifying drugs in the last month
* Intra-articular injection (hyaluronic acid/steroid) application in the last 6 months
* Having a comorbid disease that contraindicates exercise (advanced osteoporosis, vertigo, neurological diseases, etc.)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 8 weeks
  It was developed to evaluate the degree of loss of function in low back pain. Items question pain severity, self-care, lifting and carrying loads, walking, sitting, standing, sleeping, degree of pain change, travel and social life. Under each item there are six statements in which the patient ticks the one appropriate to his/her situation. The first statement is scored as "0" and the sixth statement is scored as "5". When the total score is calculated, it is multiplied by two and expressed as a percentage. The maximum score is "100" and the minimum score is "0". As the total score increases, the disability level also increases.
Y balance test | 8 weeks
  The test is a practical functional test that can predict dynamic balance and postural stability. The player's performance improves with balance, flexibility, coordination and power integration. For this test, players stand in the center of a 'Y' shaped arrangement with 3 lines drawn at certain angles. The players are asked to reach in anterior, posterolateral and posteromedial directions using one foot. Three applications are made in each direction and the average of the reach distances is recorded in centimeters. Pre-measured leg length is used to normalize the mean score of these three treatments. Percentage of maximum reach = deflection distance/leg length. Leg length; Spina iliaca anterior superior to the distal point of the medial malleolus. To obtain an overall measure of the Y Balance Test, data from all directions must be averaged to calculate the composite score.
International Physical Activity Questionnaire - Short Form | 8 weeks
  This questionnaire is a standardized tool for measuring physical activity, developed by researchers from various countries with the support of the World Health Organization (WHO) and Centers for Disease Control (CDC). Questionnaire, four areas of physical activity; It covers work, transportation, housework/gardening, and leisure activities, but also includes questions about time spent sitting as an indicator of inactivity. In each of the four areas, the energy expended in moderate and vigorous activities in the last 7 days, the number of days the activities were performed, and the number of activities performed during the day are recorded. The times are multiplied by the Metabolic Equivalent (MET) values per activity, and the results for all items are added to form the overall physical activity score. The question about sitting is not included in the physical activity score. Classification is made in three categories as physically inactive (3000 MET min/week).

CONTACTS AND LOCATIONS:
Overall Officials: Amirkiya Movahhedi, Study Chair — Bahçeşehir University
Locations (1):
- Bahçeşehir Universtiy, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Slater LV, Hart JM. Muscle Activation Patterns During Different Squat Techniques. J Strength Cond Res. 2017 Mar;31(3):667-676. doi: 10.1519/JSC.0000000000001323. PMID 26808843
- [Background] Desai I, Marshall PW. Acute effect of labile surfaces during core stability exercises in people with and without low back pain. J Electromyogr Kinesiol. 2010 Dec;20(6):1155-62. doi: 10.1016/j.jelekin.2010.08.003. PMID 20801670
- [Background] Kararti C, Ozsoy I, Ozyurt F, Basat HC, Ozsoy G, Ozudogru A. The effects of dynamic neuromuscular stabilization approach on clinical outcomes in older patients with chronic nonspecific low back pain: a randomized, controlled clinical trial. Somatosens Mot Res. 2023 Sep;40(3):116-125. doi: 10.1080/08990220.2023.2191705. Epub 2023 Mar 24. PMID 36964655